CLINICAL TRIAL: NCT01728155
Title: European Low and Intermediate Risk Neuroblastoma Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LINES
Record Dates: First submitted 2012-11-13; First posted 2012-11-16 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: LOW AND INTERMEDIATE PAEDIATRIC NEUROBLASTOMA AND NEONATAL SUPRARENAL MASSES
Keywords: NEUROBLASTOMA, LOW RISK, INTERMEDIATE RISK
MeSH Terms: conditions — Neuroblastoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Group1 (No Intervention): initial observation (chemotherapy is only given if there is subsequent progression)
- Group 1: chemotherapy (Active Comparator): chemotherapy and surgery
  Interventions: Drug: chemotherapy
- Group 2 (Experimental): chemotherapy and surgery
  Interventions: Drug: chemotherapy
- Group 3 (Experimental): chemotherapy and surgery
  Interventions: Drug: chemotherapy
- Group 4 (No Intervention): Observation
- Group 5 (Experimental): chemotherapy
  Interventions: Drug: chemotherapy
- Group 6 (Experimental): chemotherapy and surgery
  Interventions: Drug: chemotherapy
- Group 7 (Experimental): chemotherapy and surgery
  Interventions: Drug: chemotherapy
- Group 8 (Experimental): chemotherapy, surgery, radiotherapy and 13 cis-retinoic acid
  Interventions: Drug: chemotherapy
- Group 9 (Experimental): chemotherapy, surgery, radiotherapy and 13 cis-retinoic acid
  Interventions: Drug: chemotherapy
- Group 10 (Experimental): chemotherapy, surgery,
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: chemotherapy
  Arms: Group 10; Group 1: chemotherapy; Group 2; Group 3; Group 5; Group 6; Group 7; Group 8; Group 9

SUMMARY:
The European study, LINES 2009 (Low and Intermediate Risk Neuroblastoma European Study), groups together in a single protocol the treatment of all patients with "non high risk" neuroblastoma (NB), with stratification into two groups: low risk and intermediate risk. These two separate cohorts are included in one single protocol to enable patient data from these two groups to be entered into a common database, as the current prognostic classifications determining treatment may evolve further with subsequent more detailed molecular analysis of the tumours.

1. LOW RISK STUDY

The Low Risk Study is proposed in order to:

* minimise the amount of treatment (chemotherapy and surgery) for all appropriate low risk patients, who in previous studies have been shown to have an excellent long-term outcome (as in the SIOPEN 99.1-2 infant neuroblastoma studies where the overall survival was greater than 97%(H. Rubie, JCO).
* improve the EFS and maintain the OS (overall survival) in L2 and Ms patients with a SCA(Segmental Cromosomal Aberration) genomic profile tumour (presence of any segmental chromosomal change (SCA)) by electively treating these patients with chemotherapy despite the absence of symptoms.

  2) INTERMEDIATE RISK STUDY

The Intermediate Risk Study is proposed in order to:

* reduce the amount of chemotherapy for differentiating histology INRG (International Neuroblastoma Risk Group) stage L2 NB and ganglioneuroblastoma nodular patients who in previous SIOPEN study have been shown to have an excellent long-term outcome;
* increase the amount of treatment (radiotherapy and 13-cis-RA (13-cis-Retinoic Acid) for poorly differentiated or undifferentiated histology INRG stage L2 NB or ganglioneuroblastoma nodular patients in order to improve the EFS registered in the previous SIOPEN study;
* improve the EFS (Event Free Survival) of MYCN (V-Myc myelocytomatosis viral related oncogene, NB derived ,avian )amplified INSS (International NB Staging System) stage 1 NB patients with the introduction of adjuvant treatment;
* maintain the very good results obtained in previous SIOPEN study for INRG stage M infants with a moderate treatment.

NEONATAL SUPRARENAL MASSES

The incidence of suprarenal tumours/masses has increased in the last decade due to the expanded use of prenatal ultrasonography in routine obstetric care and in the neonatal and early infancy care. The differential diagnosis of these masses ranges from benign (adrenal haemorrhage) to malignant processes (neuroblastoma, adrenal carcinoma). Knowledge on perinatal suprarenal masses, although based on a relatively large literature, is scattered amongst studies on very few cases with no methodical approach and often short follow up. Therefore, the optimal management of these masses has not been clearly defined. Neuroblastoma at this age is an intriguing entity with a very good prognosis in most cases. The SIOPEN Group, based on their results in the first multicenter European Trial for infants with neuroblastoma (INES) and the world-wide experience provided in the literature, is launching this European surveillance study (Multi-centre, non-blinded, one armed prospective trial) for these masses. Treatment: Observation

DETAILED DESCRIPTION:
1. LOW RISK STUDY

The low risk group of patients includes NB patients without MYCN amplification with or without life threatening symptoms in the following clinical situations:

* Children aged ≤ 18 months with localised neuroblastoma associated with image defined risk factors precluding upfront surgery (stage INRG L2).
* Children aged ≤ 12 months with disseminated neuroblastoma without bone, pleura, lung or CNS (Central Nervous System) disease (stage INRG Ms)

  2) INTERMEDIATE RISK STUDY

The intermediate risk group of patients includes NB patients in the following clinical situations:

* Children aged >18 months with localised neuroblastoma without MYCN amplification, associated with image defined risk factors precluding upfront surgery (stage INRG L2).
* Children aged ≤12 months with disseminated neuroblastoma involving bone, pleura, lung and/or CNS (stage INRG M), without MYCN amplification.
* Children with localised resected NB (stage INSS I) with MYCN amplification. NEONATAL SUPRARENAL MASSES

The incidence of suprarenal tumours/masses has increased in the last decade due to the expanded use of prenatal ultrasonography in routine obstetric care and in the neonatal and early infancy care. The differential diagnosis of these masses ranges from benign (adrenal haemorrhage) to malignant processes (neuroblastoma, adrenal carcinoma). Knowledge on perinatal suprarenal masses, although based on a relatively large literature, is scattered amongst studies on very few cases with no methodical approach and often short follow up. Therefore, the optimal management of these masses has not been clearly defined. Neuroblastoma at this age is an intriguing entity with a very good prognosis in most cases. The SIOPEN Group, based on their results in the first multicenter European Trial for infants with neuroblastoma (INES) and the world-wide experience provided in the literature, is launching this European surveillance study (Multi-centre, non-blinded, one armed prospective trial) for these masses. Treatment: Observation

ELIGIBILITY:
1. LOW RISK STUDY

   Inclusion criteria for the whole low risk group:
   * informed consent and follow-up warranted; group assignment completed within 6 weeks from diagnosis; no prior chemotherapy or radiotherapy
   * Biopsy proven neuroblastoma
   * Tumour genomic profile obtained in a NRL according to guidelines
   * MYCN non-amplified

   Exclusion criteria for the whole low risk group:

   * Diagnosis of ganglioneuroma or ganglioneuroblastoma intermixed INRG Stage L2

   Inclusion criteria:

   *age ≤ 18 months

   Exclusion criteria:
   * any metastatic site
   * MYCN amplification
   * age > 18 months INRG Stage Ms

   Inclusion criteria:

   * age ≤ 12 months

   Exclusion criteria:
   * bone, pleura/lung and/or CNS metastasis
   * MYCN amplification
   * age > 12 months
2. INTERMEDIATE RISK STUDY

   Inclusion criteria for the whole intermediate risk group:
   * informed consent and follow-up warranted; group assignment completed within 6 weeks from diagnosis; no prior chemotherapy or radiotherapy
   * Tumour material available for biological studies according to guidelines
   * Biopsy proven neuroblastoma confirmed in a National Reference Laboratory (NRL)

   Exclusion criteria for the whole intermediate risk group:

   * Diagnosis of ganglioneuroma or ganglioneuroblastoma intermixed

   INRG Stage L1 and INSS stage 1:

   Inclusion criteria:

   * MYCN amplified

   Exclusion criteria:
   * MYCN non-amplified
   * INSS stages 2, 3, 4, 4s

   INRG Stage L2:

   Inclusion criteria:
   * Histology: differentiating, poorly differentiated, undifferentiated neuroblastoma or ganglioneuroblastoma nodular
   * MYCN non-amplified
   * age >18 months

   Exclusion criteria:
   * neuroblastoma NOS
   * MYCN amplification.
   * age ≤ 18 months

   INRG Stage M:

   Inclusion criteria:
   * Any histology
   * MYCN non-amplified
   * age ≤ 12 months

   Exclusion criteria:
   * MYCN amplification
   * age > 12 months
3. NEONATAL SUPRARENAL MASSES

Inclusion criteria:

* Age less than or equal to 90 days when the suprarenal mass is discovered.
* Suprarenal mass detected by ultrasound and/or MRI. The suprarenal mass may be cystic and/or solid, but IT CANNOT REACH THE MIDLINE AND should MEASURE ≤ 5 CM AT THE LARGEST DIAMETER.
* No regional involvement: MRI scan does not show evidence of positive ipsi/contralateral lymph nodes or other spread outside the suprarenal gland.
* No metastatic involvement.
* Frozen plasma available.
* Informed consent.
* Availability to do the adequate follow-up

Exclusion criteria:

* Age older than 90 days.
* Suprarenal mass bigger than 5 cm.
* Regional involvement.
* Metastatic involvement.
* Inability to undertake mandatory diagnostic studies (biological markers, US, MRI, MIBG).
* Follow-up not guaranteed by parents/guardians.

Ages: 90 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 685 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Primary aim for Low Risk Neuroblastoma | 2 years
  To demonstrate through a randomisation between observation and chemotherapy that you can safely reduce treatment in a subgroup of L2 low risk patients (those without life threatening symptoms (LTS) and without any segmental chromosomal changes (SCA), i.e. study group 1) by giving less treatment than has been given historically while maintaining an excellent OS of 100%.
Primary aim for Intermediate Risk Neuroblastoma | 2 years
  To improve the EFS to 70% with an OS of 90% of INRG stage L2 patients over the age of 18 months, with poorly differentiated or undifferentiated tumour histology (INPC criteria), by the addition of radiotherapy and 13-cis RA compared to historical conventional treatment (study group 8).
Primary Aim for Neonatal Suprarenal Masses | 3 year
  To maintain a 3-year event free survival over 80% with a non-operative therapeutic approach (serial monitoring, surgery if warranted) in infants with a localised suprarenal mass discovered ante or neonatally.

SECONDARY OUTCOMES:
To maintain a 2 year EFS of at least 90% and an OS of at least 95% in L2 patients with LTS without SCA (study group 2) | 2 year
To maintain the 2 year EFS of 85% and an OS of at least 98% in Ms patients without SCA (study groups 4 and 5) | 2 year
To improve the 2 year EFS to at least 90% and maintain the OS of close to 100% in L2 patients with SCA (Study Group 3) and improve the 2 year EFS to over 70% in Ms patients with SCA (study group 6) | 2 year
To evaluate adherence to the protocol recommendations regarding LTS | 5 years
To reduce surgical morbidity by promoting strict adherence to Image Defined-Risk Factors (IDRFs) to determine surgical resectability | 5 year
To define the long term follow-up and natural history of the Stage L2 non-resected masses that have remained IDRF positive at the end of treatment (study groups 1-3). | 5 year
To confirm in a larger patient cohort the excellent OS of 95% in stage M neuroblastoma without MYCN amplification, less than 12 months of age, when treated with moderate therapy (study group 10). | 3 year
Maintain the results of 3yr-EFS of 90% and 3yr-OS of 100% in stage L2 patients over the age of 18 months, with differentiating neuroblastoma or differentiating ganglioneuroblastoma nodular, despite a treatment reduction (group7) | 3 year
To improve the 3 year EFS to at least 50% and the 3 year OS to 80% in INSS stage I patients with MYCN amplified neuroblastoma by the addition of adjuvant treatment (study group 9). | 3 year
To evaluate the impact of the tumour genomic profile on patient outcome, in order to consider its role in the treatment stratification of these intermediate risk patients (all study groups). | 5 years
To manage infants with suprarenal masses discovered ante or neonatally with a uniform approach in Europe in a multicentre setting. | 5 years
To maintain an excellent overall survival with a non-operative therapeutic approach (serial monitoring, surgery if warranted) in infants with a localised suprarenal mass discovered ante or neonatally. | 3 years
To determine the 3-year surgery-free survival in infants with suprarenal masses discovered ante or neonatally and managed conservatively (non initial surgery). | 3 years
To find out the natural history of perinatal suprarenal masses, according to the definitions set up for the study. | 5 years
To study the kinetics of regression in those suspected suprarenal neuroblastomas in infants with suprarenal masses discovered ante or neonatally and managed conservatively (non initial surgery). | 5 years
To collect tissue from those suprarenal masses excised in order to perform standard and investigational pathological and biological studies (INPC, MYCN, 1p, 11). | 5 years
To collect frozen plasma from all patients included in the study in order to perform research. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Adela Cañete, MD, PhD, Study Chair — Hospital Universitari i Politècnic La Fe, Valencia, Spain; Gudrun Schleiermacher, Study Chair — Institut Curie; Kate Wheeler, Study Chair — Oxford: John Radcliffe Hospital, UK; Andrea di Cataldo, Study Chair — Policlinico Universitario, Italy; Vassilius Papadakis, Study Chair — Aghia Sophia Children's Hospital, Athens
Locations (98):
- Australia (3):
  - Monash Children's Hospital, Clayton
  - Perth Children's Hospital, Nedlands
  - Sydney Children's Hospital, Sydney
- Austria (5):
  - PHO Med Uni Graz, Graz
  - Department Kinder- und Jugendheilkunde, Innsbruck
  - Landes-Frauen- und Kinderklinik Linz, Linz
  - St. Anna Kinderspital, Vienna
  - Univ Klinik für Kinder- und Jugendheilkunde, Vienna
- Belgium (8):
  - Hôpital Universitaire d'Anvers (UZA- Universitair Ziekenhuis Antwerpen), Antwerp
  - Hôpital Universitaire des Enfants Reine Fabiola (HUDERF), Brussels
  - UCL Clíniques Universitaires Saint - Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - CHC- Clinique de l'Espérance à Liège, Liège
  - CHR de la Citadelle, Liège
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - National State Hospital (Department of Pediatrics), Copenhagen
  - University Hospital of Odense (H.C. Andersen Children´s Hospital), Odense
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Schneider Children's Medical Center, Petah Tikva
  - Ichilov Hospital Sourasky Medical Center, Tel Aviv
- Italy (29):
  - Ospedale Pediatrico G. Salesi di Ancona (Centro Regionale Oncoematologia Pediatrica), Ancona
  - Azienda Ospedaliera - Universitaria Ospedale Policlinico Consorziale, Bari
  - Azienda Ospedaliera Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliero- Universitaria di Bologna- Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale Microcitemico, Cagliari
  - Oncology Policlinico- Department of Hematology, Catania
  - Azienda Ospedaliero-Universitaria di Ferrara- Oncoematologia Pediatrica, Ferrara
  - Azienda Ospedaliero-Universitaria Ospedale Pediatrico Meyer, Florence
  - Oncology Gaslini Children's Hospital of Genova- Department of Hematology, Genova
  - Istituto Nazionale dei Tumori di Milano- Onco-ematologia Pediatrica, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena- Onco-ematologia Pediatrica, Modena
  - Azienda Ospedaliera Pediatrica Santobono Pausilipon, Napoli
  - Sec. Università degli studi di Napoli - Policlinico, Napoli
  - Azienda Ospedaliera-Universitaria di Padova- Clínica di Onco-ematologia Pediatrica, Padua
  - Ospedale dei Bambini G. Di Cristina, Palermo
  - Azienda Ospedaliero - Universitaria di Parma- Oncoematologia Pediatrica, Parma
  - Fondazione IRCCS - Policlinico San Matteo - Oncoematologia Pediadrica, Pavia
  - Azienda USL Di Pescara - U.O.C di Ematologia Clinica, Pescara
  - Ospedale Infermi di Rimini - U.O. Pediatria, Rimini
  - Ospedale Pediatrico Bambino Gesù- Oncoematologia pediatrica, Roma
  - Ospedale Policlinico Universitario Agostino Gemelli, Roma
  - Policlinico Umberto I, Roma
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Universitaria Senese - Clinica Pediatrica, Siena
  - Azienda Sanitaria Ospedaliera O.I.R.M.- Sant' Anna, Torino
  - Ospedale Cardinale G. Panico, Tricase
  - Ospedale Infantile Burlo Garofolo ( U.O. Emato-Oncologia Pediatrica - Università degli studi di Trieste), Trieste
  - Policlinico G.B. Rossi- Oncoematologia Pediatrica, Verona
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Rikshospitalet. (National coordinator), Oslo
  - University Hospital of Northern Norway, Tromsø
  - St Olavs University Hospital, Trondheim
- Spain (27):
  - Hospital de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital General Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Infanta Cristina, Badajoz
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Materno Infantil Vall d'Hebron, Barcelona
  - Hospital Universitario Cruces, Bilbao
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Materno Infantil Virgen de las Nieves, Granada
  - Hospital Materno Infantil de Jaén, Jaén
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infantil la Paz, Madrid
  - Hospital Universitario Infantil Niño Jesús, Madrid
  - Hospital Regional Universitario Carlos Haya - Hospital Materno Infantil, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Virgen del Camino, Pamplona
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto de Investigacion Sanitaria La Fe, Valencia
  - Hospital Clínic Universitari, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (6):
  - Queen Silvia's Children's Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Norrlands University Hospital, Umeå
  - Uppsala Academic Children's Hospital, Uppsala
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitäts-Kinderspital beider Basel, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - HUG Hôpitaux Universitaires Genève, Geneva
  - CHUV - Centre Hospitalier Universitaire Vaudois - Unité d'hémato-oncologie pédiatrique, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - Universitäts-Kinderspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brodeur GM, Pritchard J, Berthold F, Carlsen NL, Castel V, Castelberry RP, De Bernardi B, Evans AE, Favrot M, Hedborg F, et al. Revisions of the international criteria for neuroblastoma diagnosis, staging, and response to treatment. J Clin Oncol. 1993 Aug;11(8):1466-77. doi: 10.1200/JCO.1993.11.8.1466. PMID 8336186
- [Background] Cohn SL, Pearson AD, London WB, Monclair T, Ambros PF, Brodeur GM, Faldum A, Hero B, Iehara T, Machin D, Mosseri V, Simon T, Garaventa A, Castel V, Matthay KK; INRG Task Force. The International Neuroblastoma Risk Group (INRG) classification system: an INRG Task Force report. J Clin Oncol. 2009 Jan 10;27(2):289-97. doi: 10.1200/JCO.2008.16.6785. Epub 2008 Dec 1. PMID 19047291
- [Background] De Bernardi B, Gerrard M, Boni L, Rubie H, Canete A, Di Cataldo A, Castel V, Forjaz de Lacerda A, Ladenstein R, Ruud E, Brichard B, Couturier J, Ellershaw C, Munzer C, Bruzzi P, Michon J, Pearson AD. Excellent outcome with reduced treatment for infants with disseminated neuroblastoma without MYCN gene amplification. J Clin Oncol. 2009 Mar 1;27(7):1034-40. doi: 10.1200/JCO.2008.17.5877. Epub 2009 Jan 26. PMID 19171711
- [Background] Janoueix-Lerosey I, Schleiermacher G, Michels E, Mosseri V, Ribeiro A, Lequin D, Vermeulen J, Couturier J, Peuchmaur M, Valent A, Plantaz D, Rubie H, Valteau-Couanet D, Thomas C, Combaret V, Rousseau R, Eggert A, Michon J, Speleman F, Delattre O. Overall genomic pattern is a predictor of outcome in neuroblastoma. J Clin Oncol. 2009 Mar 1;27(7):1026-33. doi: 10.1200/JCO.2008.16.0630. Epub 2009 Jan 26. PMID 19171713
- [Background] Schleiermacher G, Michon J, Huon I, d'Enghien CD, Klijanienko J, Brisse H, Ribeiro A, Mosseri V, Rubie H, Munzer C, Thomas C, Valteau-Couanet D, Auvrignon A, Plantaz D, Delattre O, Couturier J; Societe Francaise des Cancers de l'Enfant (SFCE). Chromosomal CGH identifies patients with a higher risk of relapse in neuroblastoma without MYCN amplification. Br J Cancer. 2007 Jul 16;97(2):238-46. doi: 10.1038/sj.bjc.6603820. Epub 2007 Jun 19. PMID 17579628
- [Background] Cecchetto G, Mosseri V, De Bernardi B, Helardot P, Monclair T, Costa E, Horcher E, Neuenschwander S, Toma P, Rizzo A, Michon J, Holmes K. Surgical risk factors in primary surgery for localized neuroblastoma: the LNESG1 study of the European International Society of Pediatric Oncology Neuroblastoma Group. J Clin Oncol. 2005 Nov 20;23(33):8483-9. doi: 10.1200/JCO.2005.02.4661. PMID 16293878
- [Background] Monclair T, Brodeur GM, Ambros PF, Brisse HJ, Cecchetto G, Holmes K, Kaneko M, London WB, Matthay KK, Nuchtern JG, von Schweinitz D, Simon T, Cohn SL, Pearson AD; INRG Task Force. The International Neuroblastoma Risk Group (INRG) staging system: an INRG Task Force report. J Clin Oncol. 2009 Jan 10;27(2):298-303. doi: 10.1200/JCO.2008.16.6876. Epub 2008 Dec 1. PMID 19047290
- [Background] De Bernardi B, Mosseri V, Rubie H, Castel V, Foot A, Ladenstein R, Laureys G, Beck-Popovic M, de Lacerda AF, Pearson AD, De Kraker J, Ambros PF, de Rycke Y, Conte M, Bruzzi P, Michon J; SIOP Europe Neuroblastoma Group. Treatment of localised resectable neuroblastoma. Results of the LNESG1 study by the SIOP Europe Neuroblastoma Group. Br J Cancer. 2008 Oct 7;99(7):1027-33. doi: 10.1038/sj.bjc.6604640. Epub 2008 Sep 2. PMID 18766186
- [Background] Bagatell R, Beck-Popovic M, London WB, Zhang Y, Pearson AD, Matthay KK, Monclair T, Ambros PF, Cohn SL; International Neuroblastoma Risk Group. Significance of MYCN amplification in international neuroblastoma staging system stage 1 and 2 neuroblastoma: a report from the International Neuroblastoma Risk Group database. J Clin Oncol. 2009 Jan 20;27(3):365-70. doi: 10.1200/JCO.2008.17.9184. Epub 2008 Dec 1. PMID 19047282
- [Background] Canete A, Gerrard M, Rubie H, Castel V, Di Cataldo A, Munzer C, Ladenstein R, Brichard B, Bermudez JD, Couturier J, de Bernardi B, Pearson AJ, Michon J. Poor survival for infants with MYCN-amplified metastatic neuroblastoma despite intensified treatment: the International Society of Paediatric Oncology European Neuroblastoma Experience. J Clin Oncol. 2009 Mar 1;27(7):1014-9. doi: 10.1200/JCO.2007.14.5839. Epub 2009 Jan 26. PMID 19171715
- [Background] Hero B, Simon T, Spitz R, Ernestus K, Gnekow AK, Scheel-Walter HG, Schwabe D, Schilling FH, Benz-Bohm G, Berthold F. Localized infant neuroblastomas often show spontaneous regression: results of the prospective trials NB95-S and NB97. J Clin Oncol. 2008 Mar 20;26(9):1504-10. doi: 10.1200/JCO.2007.12.3349. PMID 18349403
- [Background] Rubie H, Michon J, Plantaz D, Peyroulet MC, Coze C, Frappaz D, Chastagner P, Baranzelli MC, Mechinaud F, Boutard P, Lutz P, Perel Y, Leverger G, de Lumley L, Millot F, Stephan JL, Margueritte G, Hartmann O. Unresectable localized neuroblastoma: improved survival after primary chemotherapy including carboplatin-etoposide. Neuroblastoma Study Group of the Societe Francaise d'Oncologie Pediatrique (SFOP). Br J Cancer. 1998 Jun;77(12):2310-7. doi: 10.1038/bjc.1998.384. PMID 9649151
- [Background] Castel V, Badal MD, Bezanilla JL, Llombart A, Ruiz-Jimenez JI, Sanchez de Toledo J, Melero C, Mulet J. Treatment of stage III neuroblastoma with emphasis on intensive induction chemotherapy: a report from the Neuroblastoma Group of the Spanish Society of Pediatric Oncology. Med Pediatr Oncol. 1995 Jan;24(1):29-35. doi: 10.1002/mpo.2950240107. PMID 7968789
- [Background] Garaventa A, De Bernardi B, Pianca C, Donfrancesco A, Cordero di Montezemolo L, Di Tullio MT, Bagnulo S, Mancini A, Carli M, Pession A, Arrighini A, Di Cataldo A, Tamaro P, Iasonni V, Taccone A, Rogers D, Boni L; Italian Cooperative Group dor Neuroblastoma. Localized but unresectable neuroblastoma: treatment and outcome of 145 cases. Italian Cooperative Group for Neuroblastoma. J Clin Oncol. 1993 Sep;11(9):1770-9. doi: 10.1200/JCO.1993.11.9.1770. PMID 8355044
- [Background] Garaventa A, Boni L, Lo Piccolo MS, Tonini GP, Gambini C, Mancini A, Tonegatti L, Carli M, di Montezemolo LC, Di Cataldo A, Casale F, Mazzocco K, Cecchetto G, Rizzo A, Bernardi B; Italian Cooperative Group for Neuroblastoma. Localized unresectable neuroblastoma: results of treatment based on clinical prognostic factors. Ann Oncol. 2002 Jun;13(6):956-64. doi: 10.1093/annonc/mdf165. PMID 12123342
- [Background] Castleberry RP, Kun LE, Shuster JJ, Altshuler G, Smith IE, Nitschke R, Wharam M, McWilliams N, Joshi V, Hayes FA. Radiotherapy improves the outlook for patients older than 1 year with Pediatric Oncology Group stage C neuroblastoma. J Clin Oncol. 1991 May;9(5):789-95. doi: 10.1200/JCO.1991.9.5.789. PMID 2016621
- [Background] Modak S, Kushner BH, LaQuaglia MP, Kramer K, Cheung NK. Management and outcome of stage 3 neuroblastoma. Eur J Cancer. 2009 Jan;45(1):90-8. doi: 10.1016/j.ejca.2008.09.016. Epub 2008 Nov 6. PMID 18996003
- [Background] Park JR, Villablanca JG, London WB, Gerbing RB, Haas-Kogan D, Adkins ES, Attiyeh EF, Maris JM, Seeger RC, Reynolds CP, Matthay KK; Children's Oncology Group. Outcome of high-risk stage 3 neuroblastoma with myeloablative therapy and 13-cis-retinoic acid: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2009 Jan;52(1):44-50. doi: 10.1002/pbc.21784. PMID 18937318
- [Background] Matthay KK, Villablanca JG, Seeger RC, Stram DO, Harris RE, Ramsay NK, Swift P, Shimada H, Black CT, Brodeur GM, Gerbing RB, Reynolds CP. Treatment of high-risk neuroblastoma with intensive chemotherapy, radiotherapy, autologous bone marrow transplantation, and 13-cis-retinoic acid. Children's Cancer Group. N Engl J Med. 1999 Oct 14;341(16):1165-73. doi: 10.1056/NEJM199910143411601. PMID 10519894
- [Background] Brodeur GM, Maris JM, Yamashiro DJ, Hogarty MD, White PS. Biology and genetics of human neuroblastomas. J Pediatr Hematol Oncol. 1997 Mar-Apr;19(2):93-101. doi: 10.1097/00043426-199703000-00001. PMID 9149737
- [Background] Maris JM, Matthay KK. Molecular biology of neuroblastoma. J Clin Oncol. 1999 Jul;17(7):2264-79. doi: 10.1200/JCO.1999.17.7.2264. PMID 10561284
- [Background] Brodeur GM. Neuroblastoma: biological insights into a clinical enigma. Nat Rev Cancer. 2003 Mar;3(3):203-16. doi: 10.1038/nrc1014. PMID 12612655
- [Background] Maris JM. The biologic basis for neuroblastoma heterogeneity and risk stratification. Curr Opin Pediatr. 2005 Feb;17(1):7-13. doi: 10.1097/01.mop.0000150631.60571.89. PMID 15659956
- [Background] Seeger RC, Brodeur GM, Sather H, Dalton A, Siegel SE, Wong KY, Hammond D. Association of multiple copies of the N-myc oncogene with rapid progression of neuroblastomas. N Engl J Med. 1985 Oct 31;313(18):1111-6. doi: 10.1056/NEJM198510313131802. PMID 4047115
- [Background] Ladenstein R, Ambros IM, Potschger U, Amann G, Urban C, Fink FM, Schmitt K, Jones R, Slociak M, Schilling F, Ritter J, Berthold F, Gadner H, Ambros PF. Prognostic significance of DNA di-tetraploidy in neuroblastoma. Med Pediatr Oncol. 2001 Jan;36(1):83-92. doi: 10.1002/1096-911X(20010101)36:13.0.CO;2-9. PMID 11464912
- [Background] Look AT, Hayes FA, Shuster JJ, Douglass EC, Castleberry RP, Bowman LC, Smith EI, Brodeur GM. Clinical relevance of tumor cell ploidy and N-myc gene amplification in childhood neuroblastoma: a Pediatric Oncology Group study. J Clin Oncol. 1991 Apr;9(4):581-91. doi: 10.1200/JCO.1991.9.4.581. PMID 2066755
- [Background] Caron H, van Sluis P, de Kraker J, Bokkerink J, Egeler M, Laureys G, Slater R, Westerveld A, Voute PA, Versteeg R. Allelic loss of chromosome 1p as a predictor of unfavorable outcome in patients with neuroblastoma. N Engl J Med. 1996 Jan 25;334(4):225-30. doi: 10.1056/NEJM199601253340404. PMID 8531999
- [Background] Luttikhuis ME, Powell JE, Rees SA, Genus T, Chughtai S, Ramani P, Mann JR, McConville CM. Neuroblastomas with chromosome 11q loss and single copy MYCN comprise a biologically distinct group of tumours with adverse prognosis. Br J Cancer. 2001 Aug 17;85(4):531-7. doi: 10.1054/bjoc.2001.1960. PMID 11506492
- [Background] Schleiermacher G, Delattre O, Peter M, Mosseri V, Delonlay P, Vielh P, Thomas G, Zucker JM, Magdelenat H, Michon J. Clinical relevance of loss heterozygosity of the short arm of chromosome 1 in neuroblastoma: a single-institution study. Int J Cancer. 1996 Apr 22;69(2):73-8. doi: 10.1002/(SICI)1097-0215(19960422)69:23.0.CO;2-S. PMID 8608986
- [Background] Attiyeh EF, London WB, Mosse YP, Wang Q, Winter C, Khazi D, McGrady PW, Seeger RC, Look AT, Shimada H, Brodeur GM, Cohn SL, Matthay KK, Maris JM; Children's Oncology Group. Chromosome 1p and 11q deletions and outcome in neuroblastoma. N Engl J Med. 2005 Nov 24;353(21):2243-53. doi: 10.1056/NEJMoa052399. PMID 16306521
- [Background] Brinkschmidt C, Christiansen H, Terpe HJ, Simon R, Lampert F, Boecker W, Dockhorn-Dworniczak B. Distal chromosome 17 gains in neuroblastomas detected by comparative genomic hybridization (CGH) are associated with a poor clinical outcome. Med Pediatr Oncol. 2001 Jan;36(1):11-3. doi: 10.1002/1096-911X(20010101)36:13.0.CO;2-M. PMID 11464859
- [Background] Lastowska M, Cullinane C, Variend S, Cotterill S, Bown N, O'Neill S, Mazzocco K, Roberts P, Nicholson J, Ellershaw C, Pearson AD, Jackson MS; United Kingdom Children Cancer Study Group and the United Kingdom Cancer Cytogenetics Group. Comprehensive genetic and histopathologic study reveals three types of neuroblastoma tumors. J Clin Oncol. 2001 Jun 15;19(12):3080-90. doi: 10.1200/JCO.2001.19.12.3080. PMID 11408505
- [Background] Plantaz D, Mohapatra G, Matthay KK, Pellarin M, Seeger RC, Feuerstein BG. Gain of chromosome 17 is the most frequent abnormality detected in neuroblastoma by comparative genomic hybridization. Am J Pathol. 1997 Jan;150(1):81-9. PMID 9006325
- [Background] Bown N, Lastowska M, Cotterill S, O'Neill S, Ellershaw C, Roberts P, Lewis I, Pearson AD; U.K. Cancer Cytogenetics Group and the U.K. Children's Cancer Study Group. 17q gain in neuroblastoma predicts adverse clinical outcome. U.K. Cancer Cytogenetics Group and the U.K. Children's Cancer Study Group. Med Pediatr Oncol. 2001 Jan;36(1):14-9. doi: 10.1002/1096-911X(20010101)36:13.0.CO;2-G. PMID 11464868
- [Background] Brinkschmidt C, Poremba C, Christiansen H, Simon R, Schafer KL, Terpe HJ, Lampert F, Boecker W, Dockhorn-Dworniczak B. Comparative genomic hybridization and telomerase activity analysis identify two biologically different groups of 4s neuroblastomas. Br J Cancer. 1998 Jun;77(12):2223-9. doi: 10.1038/bjc.1998.370. PMID 9649137
- [Background] Plantaz D, Vandesompele J, Van Roy N, Lastowska M, Bown N, Combaret V, Favrot MC, Delattre O, Michon J, Benard J, Hartmann O, Nicholson JC, Ross FM, Brinkschmidt C, Laureys G, Caron H, Matthay KK, Feuerstein BG, Speleman F. Comparative genomic hybridization (CGH) analysis of stage 4 neuroblastoma reveals high frequency of 11q deletion in tumors lacking MYCN amplification. Int J Cancer. 2001 Mar 1;91(5):680-6. doi: 10.1002/1097-0215(200002)9999:99993.0.co;2-r. PMID 11267980
- [Background] Vandesompele J, Baudis M, De Preter K, Van Roy N, Ambros P, Bown N, Brinkschmidt C, Christiansen H, Combaret V, Lastowska M, Nicholson J, O'Meara A, Plantaz D, Stallings R, Brichard B, Van den Broecke C, De Bie S, De Paepe A, Laureys G, Speleman F. Unequivocal delineation of clinicogenetic subgroups and development of a new model for improved outcome prediction in neuroblastoma. J Clin Oncol. 2005 Apr 1;23(10):2280-99. doi: 10.1200/JCO.2005.06.104. PMID 15800319
- [Background] Vandesompele J, Speleman F, Van Roy N, Laureys G, Brinskchmidt C, Christiansen H, Lampert F, Lastowska M, Bown N, Pearson A, Nicholson JC, Ross F, Combaret V, Delattre O, Feuerstein BG, Plantaz D. Multicentre analysis of patterns of DNA gains and losses in 204 neuroblastoma tumors: how many genetic subgroups are there? Med Pediatr Oncol. 2001 Jan;36(1):5-10. doi: 10.1002/1096-911X(20010101)36:13.0.CO;2-E. PMID 11464905
- [Background] Vandesompele J, Van Roy N, Van Gele M, Laureys G, Ambros P, Heimann P, Devalck C, Schuuring E, Brock P, Otten J, Gyselinck J, De Paepe A, Speleman F. Genetic heterogeneity of neuroblastoma studied by comparative genomic hybridization. Genes Chromosomes Cancer. 1998 Oct;23(2):141-52. doi: 10.1002/(sici)1098-2264(199810)23:23.0.co;2-2. PMID 9739017
- [Background] Mosse YP, Diskin SJ, Wasserman N, Rinaldi K, Attiyeh EF, Cole K, Jagannathan J, Bhambhani K, Winter C, Maris JM. Neuroblastomas have distinct genomic DNA profiles that predict clinical phenotype and regional gene expression. Genes Chromosomes Cancer. 2007 Oct;46(10):936-49. doi: 10.1002/gcc.20477. PMID 17647283
- [Background] Janoueix-Lerosey I, Hupe P, Maciorowski Z, La Rosa P, Schleiermacher G, Pierron G, Liva S, Barillot E, Delattre O. Preferential occurrence of chromosome breakpoints within early replicating regions in neuroblastoma. Cell Cycle. 2005 Dec;4(12):1842-6. doi: 10.4161/cc.4.12.2257. Epub 2005 Dec 14. PMID 16294040
- [Background] Schleiermacher G, Bourdeaut F, Combaret V, Picrron G, Raynal V, Aurias A, Ribeiro A, Janoueix-Lerosey I, Delattre O. Stepwise occurrence of a complex unbalanced translocation in neuroblastoma leading to insertion of a telomere sequence and late chromosome 17q gain. Oncogene. 2005 May 5;24(20):3377-84. doi: 10.1038/sj.onc.1208486. PMID 15735707
- [Background] Ambros IM, Benard J, Boavida M, Bown N, Caron H, Combaret V, Couturier J, Darnfors C, Delattre O, Freeman-Edward J, Gambini C, Gross N, Hattinger CM, Luegmayr A, Lunec J, Martinsson T, Mazzocco K, Navarro S, Noguera R, O'Neill S, Potschger U, Rumpler S, Speleman F, Tonini GP, Valent A, Van Roy N, Amann G, De Bernardi B, Kogner P, Ladenstein R, Michon J, Pearson AD, Ambros PF. Quality assessment of genetic markers used for therapy stratification. J Clin Oncol. 2003 Jun 1;21(11):2077-84. doi: 10.1200/JCO.2003.03.025. PMID 12775732
- [Background] Ambros PF, Ambros IM, Brodeur GM, Haber M, Khan J, Nakagawara A, Schleiermacher G, Speleman F, Spitz R, London WB, Cohn SL, Pearson AD, Maris JM. International consensus for neuroblastoma molecular diagnostics: report from the International Neuroblastoma Risk Group (INRG) Biology Committee. Br J Cancer. 2009 May 5;100(9):1471-82. doi: 10.1038/sj.bjc.6605014. PMID 19401703
- [Background] Brodeur GM, Seeger RC, Barrett A, Berthold F, Castleberry RP, D'Angio G, De Bernardi B, Evans AE, Favrot M, Freeman AI, et al. International criteria for diagnosis, staging, and response to treatment in patients with neuroblastoma. J Clin Oncol. 1988 Dec;6(12):1874-81. doi: 10.1200/JCO.1988.6.12.1874. PMID 3199170
- [Background] Shimada H, Ambros IM, Dehner LP, Hata J, Joshi VV, Roald B, Stram DO, Gerbing RB, Lukens JN, Matthay KK, Castleberry RP. The International Neuroblastoma Pathology Classification (the Shimada system). Cancer. 1999 Jul 15;86(2):364-72. PMID 10421273
- [Background] Shimada H, Ambros IM, Dehner LP, Hata J, Joshi VV, Roald B. Terminology and morphologic criteria of neuroblastic tumors: recommendations by the International Neuroblastoma Pathology Committee. Cancer. 1999 Jul 15;86(2):349-63. PMID 10421272
- [Background] Kerbl R, Urban CE, Ambros IM, Dornbusch HJ, Schwinger W, Lackner H, Ladenstein R, Strenger V, Gadner H, Ambros PF. Neuroblastoma mass screening in late infancy: insights into the biology of neuroblastic tumors. J Clin Oncol. 2003 Nov 15;21(22):4228-34. doi: 10.1200/JCO.2003.10.168. PMID 14615452
- [Background] Kerbl R, Urban CE, Lackner H, Hofler G, Ambros IM, Ratschek M, Ambros PF. Connatal localized neuroblastoma. The case to delay treatment. Cancer. 1996 Apr 1;77(7):1395-401. doi: 10.1002/(SICI)1097-0142(19960401)77:73.0.CO;2-W. PMID 8608521
- [Background] Schwab M, Westermann F, Hero B, Berthold F. Neuroblastoma: biology and molecular and chromosomal pathology. Lancet Oncol. 2003 Aug;4(8):472-80. doi: 10.1016/s1470-2045(03)01166-5. PMID 12901961
- [Background] Nadler EP, Barksdale EM. Adrenal masses in the newborn. Semin Pediatr Surg. 2000 Aug;9(3):156-64. doi: 10.1053/spsu.2000.7560. PMID 10949426
- [Background] Donoghue V, Ryan S, Twomey E. Perinatal tumours: the contribution of radiology to management. Pediatr Radiol. 2008 Jun;38 Suppl 3:S477-83. doi: 10.1007/s00247-008-0841-x. No abstract available. PMID 18470458
- [Background] Mahony R, McParland P. Approaches to the management of antenatally diagnosed congenital tumours. Pediatr Radiol. 2009 Nov;39(11):1173-8. doi: 10.1007/s00247-009-1163-3. Epub 2009 Mar 11. PMID 19277637
- [Background] Avni FE, Massez A, Cassart M. Tumours of the fetal body: a review. Pediatr Radiol. 2009 Nov;39(11):1147-57. doi: 10.1007/s00247-009-1160-6. Epub 2009 Feb 24. PMID 19238373
- [Background] Deeg KH, Bettendorf U, Hofmann V. Differential diagnosis of neonatal adrenal haemorrhage and congenital neuroblastoma by colour coded Doppler sonography and power Doppler sonography. Eur J Pediatr. 1998 Apr;157(4):294-7. doi: 10.1007/s004310050814. PMID 9578964
- [Background] Nuchtern JG. Perinatal neuroblastoma. Semin Pediatr Surg. 2006 Feb;15(1):10-6. doi: 10.1053/j.sempedsurg.2005.11.003. PMID 16458841
- [Background] Noguchi S, Masumoto K, Taguchi T, Takahashi Y, Tsuneyoshi M, Suita S. Adrenal cytomegaly: two cases detected by prenatal diagnosis. Asian J Surg. 2003 Oct;26(4):234-6. doi: 10.1016/s1015-9584(09)60312-2. PMID 14530113
- [Background] Barrette S, Bernstein ML, Leclerc JM, Champagne MA, Samson Y, Brossard J, Woods WG. Treatment complications in children diagnosed with neuroblastoma during a screening program. J Clin Oncol. 2006 Apr 1;24(10):1542-5. doi: 10.1200/JCO.2005.04.4602. PMID 16575005
- [Background] Suita S, Tajiri T, Higashi M, Tanaka S, Kinoshita Y, Takahashi Y, Tatsuta K. Insights into infant neuroblastomas based on an analysis of neuroblastomas detected by mass screening at 6 months of age in Japan. Eur J Pediatr Surg. 2007 Feb;17(1):23-8. doi: 10.1055/s-2006-924640. PMID 17407017
- [Background] Chen CP, Chen SH, Chuang CY, Lee HC, Hwu YM, Chang PY, Chen ML, Chen BF. Clinical and perinatal sonographic features of congenital adrenal cystic neuroblastoma: a case report with review of the literature. Ultrasound Obstet Gynecol. 1997 Jul;10(1):68-73. doi: 10.1046/j.1469-0705.1997.10010068.x. PMID 9263428
- [Background] Daneman A, Baunin C, Lobo E, Pracros JP, Avni F, Toi A, Metreweli C, Ho SS, Moore L. Disappearing suprarenal masses in fetuses and infants. Pediatr Radiol. 1997 Aug;27(8):675-81. doi: 10.1007/s002470050210. PMID 9252434
- [Background] Granata C, Fagnani AM, Gambini C, Boglino C, Bagnulo S, Cecchetto G, Federici S, Inserra A, Michelazzi A, Riccipetitoni G, Rizzo A, Tamaro P, Jasonni V, De Bernardi B. Features and outcome of neuroblastoma detected before birth. J Pediatr Surg. 2000 Jan;35(1):88-91. doi: 10.1016/s0022-3468(00)80020-2. PMID 10646781
- [Background] Lee SY, Chuang JH, Huang CB, Hsiao CC, Wan YL, Ng SH, Lee TY, Ko SF. Congenital bilateral cystic neuroblastoma with liver metastases and massive intracystic haemorrhage. Br J Radiol. 1998 Nov;71(851):1205-7. doi: 10.1259/bjr.71.851.10434918.
- [Background] Nishi M, Miyake H, Takeda T, Yonemori H, Hanai J, Kikuchi Y, Takasugi N. A trial to discriminate spontaneous regression from non-regression cases during mass screening for neuroblastoma. Jpn J Clin Oncol. 1994 Oct;24(5):247-51. PMID 7967103
- [Background] Wang CH, Chen SJ, Yang LY, Tang RB. Neonatal adrenal hemorrhage presenting as a multiloculated cystic mass. J Chin Med Assoc. 2008 Sep;71(9):481-4. doi: 10.1016/S1726-4901(08)70153-9. PMID 18818143
- [Background] Masiakos PT, Gerstle JT, Cheang T, Viero S, Kim PC, Wales P. Is surgery necessary for incidentally discovered adrenal masses in children? J Pediatr Surg. 2004 May;39(5):754-8. doi: 10.1016/j.jpedsurg.2004.01.039. PMID 15137013
- [Background] Oue T, Inoue M, Yoneda A, Kubota A, Okuyama H, Kawahara H, Nishikawa M, Nakayama M, Kawa K. Profile of neuroblastoma detected by mass screening, resected after observation without treatment: results of the Wait and See pilot study. J Pediatr Surg. 2005 Feb;40(2):359-63. doi: 10.1016/j.jpedsurg.2004.10.062. PMID 15750929
- [Background] Tsuchida Y, Ikeda H, Iehara T, Toyoda Y, Kawa K, Fukuzawa M. Neonatal neuroblastoma: incidence and clinical outcome. Med Pediatr Oncol. 2003 Jun;40(6):391-3. doi: 10.1002/mpo.10235. No abstract available. PMID 12692810
- [Background] Sauvat F, Sarnacki S, Brisse H, Medioni J, Rubie H, Aigrain Y, Gauthier F, Audry G, Helardot P, Landais P, Michon J, Hartmann O, Nihoul-Fekete C. Outcome of suprarenal localized masses diagnosed during the perinatal period: a retrospective multicenter study. Cancer. 2002 May 1;94(9):2474-80. doi: 10.1002/cncr.10502. PMID 12015773
- [Background] Crofton PM, Squires N, Davidson DF, Henderson P, Taheri S. Reliability of urine collection pads for routine and metabolic biochemistry in infants and young children. Eur J Pediatr. 2008 Nov;167(11):1313-9. doi: 10.1007/s00431-008-0733-y. Epub 2008 May 21. PMID 18493793
- [Background] Kellie SJ, Clague AE, McGeary HM, Smith PJ. The value of catecholamine metabolite determination on untimed urine collections in the diagnosis of neural crest tumours in children. Aust Paediatr J. 1986 Nov;22(4):313-5. doi: 10.1111/j.1440-1754.1986.tb02156.x. PMID 3566681
- [Background] Pussard E, Neveux M, Guigueno N. Reference intervals for urinary catecholamines and metabolites from birth to adulthood. Clin Biochem. 2009 Apr;42(6):536-9. doi: 10.1016/j.clinbiochem.2008.10.022. Epub 2008 Nov 11. PMID 19027729
- [Background] Snow AB, Khalyfa A, Serpero LD, Capdevila OS, Kim J, Buazza MO, Gozal D. Catecholamine alterations in pediatric obstructive sleep apnea: effect of obesity. Pediatr Pulmonol. 2009 Jun;44(6):559-67. doi: 10.1002/ppul.21015. PMID 19431192
- [Background] Combaret V, Audoynaud C, Iacono I, Favrot MC, Schell M, Bergeron C, Puisieux A. Circulating MYCN DNA as a tumor-specific marker in neuroblastoma patients. Cancer Res. 2002 Jul 1;62(13):3646-8. PMID 12097268
- [Background] Gotoh T, Hosoi H, Iehara T, Kuwahara Y, Osone S, Tsuchiya K, Ohira M, Nakagawara A, Kuroda H, Sugimoto T. Prediction of MYCN amplification in neuroblastoma using serum DNA and real-time quantitative polymerase chain reaction. J Clin Oncol. 2005 Aug 1;23(22):5205-10. doi: 10.1200/JCO.2005.02.014. PMID 16051962
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Ambros PF, Ambros IM, Kerbl R, Luegmayr A, Rumpler S, Ladenstein R, Amann G, Kovar H, Horcher E, De Bernardi B, Michon J, Gadner H. Intratumoural heterogeneity of 1p deletions and MYCN amplification in neuroblastomas. Med Pediatr Oncol. 2001 Jan;36(1):1-4. doi: 10.1002/1096-911X(20010101)36:13.0.CO;2-L. PMID 11464855
- [Background] Stark DD, Moss AA, Brasch RC, deLorimier AA, Albin AR, London DA, Gooding CA. Neuroblastoma: diagnostic imaging and staging. Radiology. 1983 Jul;148(1):101-5. doi: 10.1148/radiology.148.1.6856817.
- [Background] Brody AS, Frush DP, Huda W, Brent RL; American Academy of Pediatrics Section on Radiology. Radiation risk to children from computed tomography. Pediatrics. 2007 Sep;120(3):677-82. doi: 10.1542/peds.2007-1910. PMID 17766543
- [Background] Semelka RC, Armao DM, Elias J Jr, Huda W. Imaging strategies to reduce the risk of radiation in CT studies, including selective substitution with MRI. J Magn Reson Imaging. 2007 May;25(5):900-9. doi: 10.1002/jmri.20895. PMID 17457809
- [Background] Siegel MJ, Jaju A. MR imaging of neuroblastic masses. Magn Reson Imaging Clin N Am. 2008 Aug;16(3):499-513, vi. doi: 10.1016/j.mric.2008.04.007. PMID 18585601
- [Background] Sofka CM, Semelka RC, Kelekis NL, Worawattanakul S, Chung CJ, Gold S, Fordham LA. Magnetic resonance imaging of neuroblastoma using current techniques. Magn Reson Imaging. 1999 Feb;17(2):193-8. doi: 10.1016/s0730-725x(98)00102-7. PMID 10215473
- [Background] Lonergan GJ, Schwab CM, Suarez ES, Carlson CL. Neuroblastoma, ganglioneuroblastoma, and ganglioneuroma: radiologic-pathologic correlation. Radiographics. 2002 Jul-Aug;22(4):911-34. doi: 10.1148/radiographics.22.4.g02jl15911. PMID 12110723
- [Background] Brisse HJ, Aubert B. [CT exposure from pediatric MDCT: results from the 2007-2008 SFIPP/ISRN survey]. J Radiol. 2009 Feb;90(2):207-15. doi: 10.1016/s0221-0363(09)72471-0. French. PMID 19308005
- [Background] Goske MJ, Applegate KE, Boylan J, Butler PF, Callahan MJ, Coley BD, Farley S, Frush DP, Hernanz-Schulman M, Jaramillo D, Johnson ND, Kaste SC, Morrison G, Strauss KJ, Tuggle N. The Image Gently campaign: working together to change practice. AJR Am J Roentgenol. 2008 Feb;190(2):273-4. doi: 10.2214/AJR.07.3526. No abstract available. PMID 18212208
- [Background] Boglino C, Martins AG, Ciprandi G, Sousinha M, Inserra A. Spinal cord vascular injuries following surgery of advanced thoracic neuroblastoma: an unusual catastrophic complication. Med Pediatr Oncol. 1999 May;32(5):349-52. doi: 10.1002/(sici)1096-911x(199905)32:53.0.co;2-p. PMID 10219336
- [Background] Ou P, Schmit P, Layouss W, Sidi D, Bonnet D, Brunelle F. CT angiography of the artery of Adamkiewicz with 64-section technology: first experience in children. AJNR Am J Neuroradiol. 2007 Feb;28(2):216-9. PMID 17296982
- [Background] Goo HW, Choi SH, Ghim T, Moon HN, Seo JJ. Whole-body MRI of paediatric malignant tumours: comparison with conventional oncological imaging methods. Pediatr Radiol. 2005 Aug;35(8):766-73. doi: 10.1007/s00247-005-1459-x. Epub 2005 Apr 28. PMID 15864576
- [Background] Uhl M, Altehoefer C, Kontny U, Il'yasov K, Buchert M, Langer M. MRI-diffusion imaging of neuroblastomas: first results and correlation to histology. Eur Radiol. 2002 Sep;12(9):2335-8. doi: 10.1007/s00330-002-1310-9. Epub 2002 Mar 19. PMID 12195491
- [Background] Mendichovszky IA, Marks SD, Simcock CM, Olsen OE. Gadolinium and nephrogenic systemic fibrosis: time to tighten practice. Pediatr Radiol. 2008 May;38(5):489-96; quiz 602-3. doi: 10.1007/s00247-007-0633-8. Epub 2007 Oct 18. PMID 17943276
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Lumbroso J, Guermazi F, Hartmann O, Coornaert S, Rabarison Y, Lemerle J, Parmentier C. [Sensitivity and specificity of meta-iodobenzylguanidine (mIBG) scintigraphy in the evaluation of neuroblastoma: analysis of 115 cases]. Bull Cancer. 1988;75(1):97-106. French. PMID 3359060
- [Background] Khafagi FA, Shapiro B, Fischer M, Sisson JC, Hutchinson R, Beierwaltes WH. Phaeochromocytoma and functioning paraganglioma in childhood and adolescence: role of iodine 131 metaiodobenzylguanidine. Eur J Nucl Med. 1991;18(3):191-8. doi: 10.1007/BF02262730. PMID 1645665
- [Background] Leung A, Shapiro B, Hattner R, Kim E, de Kraker J, Ghazzar N, Hartmann O, Hoefnagel CA, Jamadar DA, Kloos R, Lizotte P, Lumbroso J, Rufini V, Shulkin BL, Sisson JC, Thein A, Troncone L. Specificity of radioiodinated MIBG for neural crest tumors in childhood. J Nucl Med. 1997 Sep;38(9):1352-7. PMID 9293786
- [Background] Shapiro B, Copp JE, Sisson JC, Eyre PL, Wallis J, Beierwaltes WH. Iodine-131 metaiodobenzylguanidine for the locating of suspected pheochromocytoma: experience in 400 cases. J Nucl Med. 1985 Jun;26(6):576-85. PMID 2860214
- [Background] Shulkin BL, Shapiro B. Current concepts on the diagnostic use of MIBG in children. J Nucl Med. 1998 Apr;39(4):679-88. PMID 9544682
- [Background] Sisson JC, Shulkin BL. Nuclear medicine imaging of pheochromocytoma and neuroblastoma. Q J Nucl Med. 1999 Sep;43(3):217-23. PMID 10568137
- [Background] Wieland DM, Wu J, Brown LE, Mangner TJ, Swanson DP, Beierwaltes WH. Radiolabeled adrenergi neuron-blocking agents: adrenomedullary imaging with [131I]iodobenzylguanidine. J Nucl Med. 1980 Apr;21(4):349-53. PMID 7381563
- [Background] Khafagi FA, Shapiro B, Gross MD. The adrenal gland. In: Maisey MN, Britton KE, Gilday DL, eds. Clinical Nuclear Medicine. 2nd ed: London Chapman & Hall 1989:271-91.
- [Background] Wilson LM, Draper GJ. Neuroblastoma, its natural history and prognosis: a study of 487 cases. Br Med J. 1974 Aug 3;3(5926):301-7. doi: 10.1136/bmj.3.5926.301. PMID 4414795
- [Background] Young JL Jr, Ries LG, Silverberg E, Horm JW, Miller RW. Cancer incidence, survival, and mortality for children younger than age 15 years. Cancer. 1986 Jul 15;58(2 Suppl):598-602. doi: 10.1002/1097-0142(19860715)58:2+3.0.co;2-c. PMID 3719551
- [Background] Gelfand MJ. Meta-iodobenzylguanidine in children. Semin Nucl Med. 1993 Jul;23(3):231-42. doi: 10.1016/s0001-2998(05)80104-7. PMID 8378796
- [Background] Jacobs A, Delree M, Desprechins B, Otten J, Ferster A, Jonckheer MH, Mertens J, Ham HR, Piepsz A. Consolidating the role of *I-MIBG-scintigraphy in childhood neuroblastoma: five years of clinical experience. Pediatr Radiol. 1990;20(3):157-9. doi: 10.1007/BF02012960. PMID 2352793
- [Background] Lumbroso JD, Guermazi F, Hartmann O, Coornaert S, Rabarison Y, Leclere JG, Couanet D, Bayle C, Caillaud JM, Lemerle J, et al. Meta-iodobenzylguanidine (mIBG) scans in neuroblastoma: sensitivity and specificity, a review of 115 scans. Prog Clin Biol Res. 1988;271:689-705. No abstract available. PMID 3261424
- [Background] Parisi MT, Greene MK, Dykes TM, Moraldo TV, Sandler ED, Hattner RS. Efficacy of metaiodobenzylguanidine as a scintigraphic agent for the detection of neuroblastoma. Invest Radiol. 1992 Oct;27(10):768-73. doi: 10.1097/00004424-199210000-00003. PMID 1399431
- [Background] Perel Y, Conway J, Kletzel M, Goldman J, Weiss S, Feyler A, Cohn SL. Clinical impact and prognostic value of metaiodobenzylguanidine imaging in children with metastatic neuroblastoma. J Pediatr Hematol Oncol. 1999 Jan-Feb;21(1):13-8. doi: 10.1097/00043426-199901000-00004. PMID 10029806
- [Background] Moyes J, McCready VR, Fullbrook AC. Neuroblastoma MIBG in its diagnosis and management: Springer-Verlag Berlin and Heidelberg GmbH & Co. K 1989.
- [Background] Hoefnagel CA, De Kraker J, Valdes Olmos RA, Voute PA. [131I]MIBG as a first line treatment in advanced neuroblastoma. Q J Nucl Med. 1995 Dec;39(4 Suppl 1):61-4. PMID 9002752
- [Background] Lumbroso J, Hartmann O, Schlumberger M. Therapeutic use of [131I]metaiodobenzylguanidine in neuroblastoma: a phase II study in 26 patients. "Societe Francaise d'Oncologie Pediatrique" and Nuclear Medicine Co-investigators. J Nucl Biol Med (1991). 1991 Oct-Dec;35(4):220-3. PMID 1823822
- [Background] Mairs RJ. Neuroblastoma therapy using radiolabelled [131I]meta-iodobenzylguanidine ([131I]MIBG) in combination with other agents. Eur J Cancer. 1999 Aug;35(8):1171-3. doi: 10.1016/s0959-8049(99)00114-8. No abstract available. PMID 10615225
- [Background] Gordon I, Peters AM, Gutman A, Morony S, Dicks-Mireaux C, Pritchard J. Skeletal assessment in neuroblastoma--the pitfalls of iodine-123-MIBG scans. J Nucl Med. 1990 Feb;31(2):129-34. PMID 2313350
- See also: The European Network for Cancer Research in Children and Adolescents (ENCCA) is a Network of Excellence Funded by the European Union's 7th Framework Programme (FP7): See WP10 — https://www.siope.eu/activities/eu-projects/encca/